CLINICAL TRIAL: NCT01162278
Title: Dose Escalating Study of Single Fraction Stereotactic Body Radiation Therapy (SBRT) for Patients With Hepatic Metastases
Brief Title: Stereotactic Body Radiation Therapy (SBRT) for Patients With Hepatic Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 072010-093
Record Dates: First submitted 2010-06-25; First posted 2010-07-14 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2018-01

CONDITIONS: Liver Metastases
Keywords: liver metastases; Stereotactic Body Radiation Therapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single fraction (Other): Patients in each dose cohort will all be treated as a single group for dose escalation. The starting dose for the dose escalation portion will be 35Gy in one fraction. Subsequent cohorts of patients will receive an additional 5Gy per treatment to a maximum planned dose of 50Gy in one fraction.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Single fraction SBRT
  Other Names: Stereotactic Body Radiation Therapy

SUMMARY:
Patients that have had staging studies identifying them as AJCC stage IV with up to five liver metastases will be considered for the study. About 60 patients will take part in this study at UT southwestern, Parkland Health & Hospital System, and Methodist Richardson Cancer Center. There are four dose cohorts for this study and each cohort will enroll a minimum of 7 to a maximum of 15 patients depending on tolerance of therapy. The treatment period will last for approximately 1 day and the follow-up portion of the study will last 5 years.

DETAILED DESCRIPTION:
If the patient has met all the eligibility criteria, they will be registered to the study After successful registration to the study and treatment planning session, patients will receive a single fraction of radiation. The total dose a particular patient receives will depend on the dose cohort they are enrolled into. Each treatment will last about one hour and will be given in a particular position to help guide the beams of radiation toward the cancer area. Although it is not mandatory, it is recommended that patients receive corticosteroid premedication (e.g. Decadron 4-10 m.g. p.o. in a single dose or equivalent) 15-60 minutes prior to each treatment for the intended purpose of modulating immediate acute inflammatory effects and providing anti-emetic support.

ELIGIBILITY:
Inclusion Criteria:

* Signed study specific informed consent form.
* Age ≥ 18.
* Zubrod Performance Status 0-2.
* Biopsy proven primary malignancy.
* Predicted survival of >6 months.
* AJCC Stage IV disease with up to 5 liver metastases as seen on a contrast- enhanced CT, MRI or PET/CT.
* Ability to spare a critical liver volume as defined by the protocol constraints.
* Tumors must be located outside the Central Liver Zone defined by contouring the portal vein to its bifurcation + a 3-dimensional 2cm margin

Exclusion Criteria:

* Patients with a history of prior irradiation or other treatment to the liver or abdomen who after the protocol treatment would have cumulative doses to the liver or other normal tissues greater than the protocol defined constraints.
* Need or plans for concomitant antineoplastic therapy (including surgery, cryotherapy, radiofrequency ablation, chemo-embolization, conventionally fractionated radiotherapy, brachytherapy, and hepatic artery chemotherapy) for the protocol treated lesions except at progression. Adjuvant systemic therapy before and after the protocol therapy per section 7.0, and surgery or other ablative therapy is allowed for lesions appearing after enrollment to this protocol as per section 8.0 is allowed.
* Germ cell or hematologic malignancies.
* History of Crohn's Disease or Ulcerative Colitis.
* Active peptic ulcer disease.
* Underlying hepatic cirrhosis with Child-Pugh class B or C
* A major psychiatric illness which would limit understanding of the proposed protocol treatment and consent process
* Men and women of reproductive potential may not participate unless they agree to use an effective contraceptive method.
* Pregnant or lactating women.
* Severe, active co-morbidity
* Abnormal labs

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-07 (Actual); Primary Completion 2015-11-25 (Actual); Study Completion 2017-11-25 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose of single fraction stereotactic radiotherapy in patients with hepatic metastases. | 3 years
  The dose of single fraction stereotactic radiotherapy will be escalated without exceeding the maximum tolerated dose in patients with hepatic metastases.

SECONDARY OUTCOMES:
The dose-limiting toxicity. | 3 years
The actual 6 and 12 month local control rates | 4 years
An optimal therapeutic window between control and toxicity | 3 years
The 3 month tumor response rate | 3 month
The survival rate | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States